CLINICAL TRIAL: NCT04535076
Title: Cognitive Outcome After Surgical and Transcatheter Aortic Valve Replacement
Acronym: COSTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heart and Brain Research Group, Germany (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MC 68/2017
Record Dates: First submitted 2020-08-27; First posted 2020-09-01 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2022-03

CONDITIONS: Postoperative Delirium; Postoperative Cognitive Dysfunction; Transcatheter Aortic Valve Replacement; Surgical Aortic Valve Replacement
MeSH Terms: conditions — Emergence Delirium; Postoperative Cognitive Complications | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcatheter Aortic Valve Implantation (Experimental)
  Interventions: Procedure: Transcatheter Aortic Valve Implantation
- Surgical Aortic Valve Replacement (Active Comparator)
  Interventions: Procedure: Surgical Aortic Valve Replacement

INTERVENTIONS:
Procedure: Transcatheter Aortic Valve Implantation — Transcatheter Aortic Valve Implantation
  Arms: Transcatheter Aortic Valve Implantation
Procedure: Surgical Aortic Valve Replacement — Surgical Aortic Valve Replacement
  Arms: Surgical Aortic Valve Replacement

SUMMARY:
Aortic valve stenosis is one of the most common types of heart disease in the aging Western population. While surgical cardiac valve replacement (SAVR) is a standard therapy for patients with aortic stenosis, catheter-assisted aortic valve implantation (TAVI) has developed as an alternative to open-heart surgery, especially for high-risk patients. Recently, increased surgeon experience and improved transcatheter valve systems have led to a global trend to use TAVI in patients with low or intermediate risk. Although cognitive impairment after cardiac surgery is well known, the effect of TAVI on cognitive function has not yet been adequately investigated. The aim of this study is to compare the occurrence and progression of delirium, postoperative cognitive decline (POCD), cerebral infarction, and health-related quality of life (QOL) in patients with intermediate risk for catheter-assisted (TAVI) and surgical (SAVR) aortic valve replacement.

DETAILED DESCRIPTION:
The present project is a substudy of the DEDICATE Trial (ID: NCT03112980). It is a randomized intervention study taking place at the Kerckhoff-Klink Bad Nauheim Germany (Campus Justus Liebig University Giessen) involving 100 patients undergoing aortic valve replacement (TAVI vs. SAVR) with a focus on cognitive outcome. A detailed assessment of psychological and health-related functions will be performed before intervention, during hospitalization and 3 months after intervention. During hospitalization, the occurrence and progression of delirium will be assessed with the Intensive Care Delirium Screening Checklist (ICDSC). Other cognitive data will be collected before and 3 months after surgery with a selected and comprehensive neuropsychological test battery, including the evaluation of attention, word fluency, executive functions and various functional areas of memory. In addition, parameters of health-related QOL will be collected before and 3 months after the intervention using the SF-36, and information on anxiety and depression will be collected using the Hospital Anxiety and Depression Scale (HADS). A few days after the intervention, magnetic resonance images of the brain will be acquired to assess cerebral infarction.

ELIGIBILITY:
Inclusion Criteria:

1. Heart team decision that both TAVI and SAVR are medically justified based on

   * Degenerative aortic valve stenosis:

     * Mean gradient > 40 mmHg or
     * Jet velocity > 40 m/s or
     * Surface of aortic valve < 1.0 cm²
   * Patient shows symptoms of aortic stenosis

     * NYHA functional class ≥ II or
     * Angina pectoris or
     * Syncope
   * Low to intermediate surgical risk (STS: 2-6%)
   * A transfemoral or alternative access for TAVI can be implemented
2. Patient has agreed in writing to participate in the study
3. Patient is able to understand the patient information and sign it personally
4. Patient agrees to undergo SAVR if randomization into the control group occurs
5. Readiness for MRT examination and neuropsychological testing after 3 months
6. Patients aged 65 to 85 years.
7. Native German speaker (since a neuropsychological test is language dependent)

Exclusion Criteria:

1. Congenital aortic valve defects
2. Untreated clinically significant coronary artery disease or severe mitral or tricuspid insufficiency or mitral stenosis
3. Previous heart surgery
4. Percutaneous coronary intervention performed within one month prior to the study
5. Hemodynamic instability requiring inotropic support or mechanical circulatory support
6. Ischemic stroke or intracranial bleeding within the month before the start of the study
7. Severe ventricular dysfunction with left ventricular ejection fraction < 20% as measured by echocardiogram
8. Hypertrophic obstructive cardiomyopathy or severe basal septum hypertrophy
9. Echocardiographic detection of intracardiac mass, thrombus, vegetation, or endocarditis
10. Any other atherosclerotic disease that is considered as a contraindication for isolated aortic valve surgery
11. Symptomatic carotid or vertebral artery disease
12. Existing neurological or psychiatric disease (particularly cerebral infarction, cranio- cerebral trauma, manifest depression or dementia) that may interfere with neuropsychological testing.
13. Contraindications for MRI examination (e.g. cardiac pacemaker, vena cava filter, claustrophobia)

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2022-12-19 (Actual)

PRIMARY OUTCOMES:
Number of participants with postoperative cognitive decline at 3 months after surgery, defined as a decrease between pre- and postoperative examinations of one standard deviation in at least 20% of all objective neuropsychological parameters | Immediately pre-surgery to 3 months post-surgery
  The objective neuropsychological parameters measure cognitive domains like immediate memory span, free recall, recognition memory, selective attention, working memory, inhibition and word fluency. These cognitive domains will be measured with the following instruments: "Verbaler Lern- und Merkfähigkeitstest" (VLMT), "Trail Making Test A/B" (TMT), "Letter Number Span Test" (LNS), Block Tapping Test (BTT), "Regensburger Wortflüssigkeits-Test" (RWT), and "Syndrom-Kurz Test" (SKT).
Number of participants with postoperative cognitive decline at the time of discharge from the acute clinic, defined as a decrease between the pre- and postoperative examinations of one standard deviation measured with the "Montreal Cognitive Assessment" | Immediately pre-surgery to approximately 1 week post-surgery
  The "Montreal Cognitive Assessment" (MOCA) is a screening procedure for general cognitive function.
Number of participants with postoperative delirium during the stay in the intensive care unit as assessed by the "Intensive Care Delirium Screening Checklist" (ICDSC) | Immediately post-surgery to approximately 7 days post-surgery
  Postoperative delirium is defined as the occurrence of at least one delirious episode during a stay in the intensive care unit. The "Intensive Care Delirium Screening Checklist" (ICDSC) record the clinical symptoms of consciousness, attention, orientation, hallucinations, psychomotor retardation or agitation, speech, and changing symptoms by observing behavior and asking concrete questions to the patient.

SECONDARY OUTCOMES:
Change from baseline cognitive failures in everyday life at 3 months after surgery as assessed by the "Cognitive Failures Questionnaire" (CFQ) | Immediately pre-surgery to 3 months post-surgery
  The "Cognitive Failures Questionnaire" (CFQ) measure the frequency of failures in daily living in terms of memory, attention, action, and perception. It comprises 29 questions, which are answered on a 5-step Likert scale. Higher scores mean a worse outcome.
Change from baseline health-related quality of life at 3 months after surgery as assessed by the "36-Item Short Form Health Survey" (SF36) | Immediately pre-surgery to 3 months post-surgery
  The "36-Item Short Form Health Survey" (SF36) includes 36 questions covering 8 health-related factors: vitality, physical functioning, bodily pain, general health perception, physical role function, emotional role function, social role functioning, and mental health. An aggregated percentage score is calculated for each of the eight factors. The percentage scores range from 0% to 100%. Higher scores mean a better outcome.
Change from baseline anxiety at 3 months after surgery as assessed by the "Hospital Anxiety and Depression Scale" (HADS). | Immediately pre-surgery to 3 months post-surgery
  With the "Hospital Anxiety and Depression Scale" (HADS), an instrument will be used that refers to the psychological core aspects of depression and anxiety. Each scale contains 7 questions to be answered on a 4-step Likert scale by the patients themselves. After inverting negative questions, higher scores mean a worse outcome.
Change from baseline depression at 3 months after surgery as assessed by the "Hospital Anxiety and Depression Scale" (HADS). | Immediately pre-surgery to 3 months post-surgery
  With the "Hospital Anxiety and Depression Scale" (HADS), an instrument will be used that refers to the psychological core aspects of depression and anxiety. Each scale contains 7 questions to be answered on a 4-step Likert scale by the patients themselves. After inverting negative questions, higher scores mean a worse outcome.
Number of participants with postoperative acute ischemic lesions at the time of discharge from the acute clinic as assessed by magnetic resonance images (MRI). | Once within the 6th-10th day immediately post-surgery
  Cranial MRI will be performed using a 3-T scanner (Skyra; Siemens, Erlangen, Germany). The protocol of imaging will include a T2-weighted turbo spin-echo sequence, a T2-weighted turbo spin-echo sequence for dark fluid, a T1-weighted FLASH sequence and a diffusion-weighted echo-planar imaging sequence.
Number of participants with postoperative microemboli at the time of discharge from the acute clinic as assessed by magnetic resonance images (MRI). | Once within the 6th-10th day immediately post-surgery
  Cranial MRI will be performed using a 3-T scanner (Skyra; Siemens, Erlangen, Germany). The protocol of imaging will include a T2-weighted turbo spin-echo sequence, a T2-weighted turbo spin-echo sequence for dark fluid, a T1-weighted FLASH sequence and a diffusion-weighted echo-planar imaging sequence.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Jünemann, Dr.med.M.Sc., Principal Investigator — Clinic for Neurology, University Hospital Giessen; Marius Butz, Dipl.-Psych., Principal Investigator — Department of Cardiac Surgery, Kerckhoff Clinic Bad Nauheim; Tibo Gerriets, Prof.Dr.med., Principal Investigator — Department of Neurology, Gesundheitszentrum Wetterau; Markus Schönburg, Prof.Dr.med., Principal Investigator — Department of Cardiac Surgery, Kerckhoff Clinic Bad Nauheim; Won-Keun Kim, Dr.med., Principal Investigator — Department of Cardiac Surgery, Kerckhoff Clinic Bad Nauheim
Locations (1):
- Department of Cardiac Surgery, Kerckhoff-Klinik GmbH, Bad Nauheim, Germany

REFERENCES:
- [Derived] Butz M, Juenemann M, El-Shazly J, Meyer R, Gerriets T, Braun T, Yenigun M, Schmidt H, Tschernatsch M, Schramm P, Alhaj-Omar O, Kirchhof A, Choi YH, Sossalla S, Renker M, Blankenberg S, Seiffert M, Schoenburg M, Kim WK. Neurocognition and health-related quality of life in patients randomized to surgical or transcatheter aortic-valve replacement. Clin Res Cardiol. 2026 Feb 5. doi: 10.1007/s00392-026-02862-1. Online ahead of print. PMID 41642336